CLINICAL TRIAL: NCT03011944
Title: Assessing the Impact of a Comprehensive Nutrition-Focused Quality Improvement Program (QIP) on Health and Economic Outcomes of Malnourished Adult Patients Across the Continuum of Care
Brief Title: Impact of a Nutrition Quality Improvement Program on Outcomes of Malnourished Patients
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: HA25
Record Dates: First submitted 2016-12-28; First posted 2017-01-06 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Quality Improvement Program: This group will consist of hospitalized and SNF, at-risk/malnourished patients being discharged to home health and outpatients at-risk/malnourished patients enrolled in home health.
  Interventions: Other: Quality Improvement Program
- Control: This group will consist of historical controls, concurrent controls, and matched concurrent controls across other sites within the health system.

INTERVENTIONS:
Other: Quality Improvement Program — Nutrition screening, Nutrition consult, Oral Nutritional Supplement will be implemented in the Home Health branches as standard of care.
  Groups: Quality Improvement Program

SUMMARY:
A nutrition-focused QIP will be implemented as standard of care at select branches of the home health division of the health care system. The QIP will be comprised of three groups of patients, Group 1 will consist of hospitalized, at-risk/malnourished patients being discharged to home health, Group 2 will consist of outpatients at-risk/malnourished patients enrolled in home health and Group 3 will consist of SNF, at-risk/malnourished patients being discharged to home health. Groups will be followed for 90 days post enrollment. The QIP groups will be compared to historical controls, concurrent controls, and matched concurrent controls across other sites within the health system.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to home health from within the healthcare system's hospitals, skilled nursing facility (SNF) or outpatient clinics
* Patient is screened positive for malnutrition during hospital stay and/or by home health nutrition screening tool upon enrollment into home health
* Patient is able to consume foods and beverages orally and the physician has not indicated otherwise

Exclusion Criteria:

* Enrollment to home health from a hospital, SNF or outpatient clinic not affiliated with the healthcare system
* Patient is pregnant
* Patient is intubated, receiving tube feeding or parenteral nutrition
* Patient has severe dementia or delirium
* History of significant psychiatric disorder
* Any other disorder that may interfere with QIP product consumption or compliance with QIP protocol procedures as per the admitting clinicians
* Subject has stated an allergy or intolerance to any of the ONS ingredients
* Patients receiving hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malnourished patients receiving care in the targeted branch of the home health division of the health care system.
Sampling Method: Non-Probability Sample
Enrollment: 1546 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Hospital readmissions or admissions | Enrollment to Home Health to 90 Days

SECONDARY OUTCOMES:
Healthcare resource utilization and costs | Enrollment to Home Health to 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Suela Sulo, PhD, MSc, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Advocate at Home, Des Plaines, Illinois
  - Advocate at Home- South Office, Oak Lawn, Illinois

IPD SHARING:
Plan to Share IPD: Undecided